CLINICAL TRIAL: NCT01113437
Title: The Effect of a Humanised Monoclonal Anti-IgE Antibody,Omalizumab, on Disease Control and Bronchial Mucosal Inflammation in Non-atpic Asthma
Brief Title: Omalizumab in Non-atopic Asthma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Prof. Christopher Corrigan, King's College, London, United Kingdom
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09/H0804/43; 2009-009154-25 (EudraCT Number)
Record Dates: First submitted 2010-04-26; First posted 2010-04-29 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2010-04

CONDITIONS: Bronchial Asthma
Keywords: Bronchial Asthma; Allergy
MeSH Terms: conditions — Asthma; Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omalizumab (Experimental): There are 2 arms of the study; patients in one arm receiving omalizumab and in the other arm receiving placebo.
  Interventions: Drug: Omalizumab
- Placebo (Placebo Comparator): There are 2 arms of the study; patients in one arm receiving omalizumab and in the other arm receiving placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omalizumab — Omalizumab or placebo by subcutaneous injections, at 4 weekly or 2 weekly intervals.
  Dosage is according to manufacturer's guidance and calculated based on body weight and total serum IgE.
  Other Names: Xolair
  Arms: Omalizumab
Drug: Placebo — Omalizumab or placebo by subcutaneous injections, at 4 weekly or 2 weekly intervals.
  Dosage is according to manufacturer's guidance and calculated based on body weight and total serum IgE.
  Arms: Placebo

SUMMARY:
Hypothesis- Omalizumab(humanized monoclonal anti-IgE antibody)improves disease control and reduces bronchial mucosal inflammation in non-atopic asthma.

In order to test the above hypothesis, the investigators propose a placebo controlled, double blind, parallel group study to obtain proof of principle that omalizumab exerts beneficial effects on disease control in non-atopic severe adult asthmatics aged 18-60 years . Forty patients will be randomized in a 1:1 ratio to receive omalizumab or matching placebo. Following 12 weeks of treatment with omalizumab/placebo, and as this treatment is continued for a further 8 weeks, anti-asthma treatment will be reduced. Dosages will be administered at 4 or 2 weekly intervals over a 16 week period (5 or 10 doses in total), which corresponds with the time stated as necessary to judge efficacy of therapy according to omalizumab's licensed indications in atopic asthma. Efficacy will be judged by clinical monitoring and by bronchial biopsy to assess effects on bronchial inflammation and local IgE production.

DETAILED DESCRIPTION:
The primary aim of the study is to obtain proof of principle that omalizumab therapy maintains lung function, symptom control and quality of life in a group of non-atopic, moderate/severe asthmatics whose regular anti-asthma therapy is uniformised and reduced for an 8 week period following omalizumab/placebo therapy while the latter therapy is continued.

A secondary aim is to see whether omalizumab, as compared with placebo therapy reduces bronchial inflammation and local IgE production in the bronchial mucosa of this same group of asthmatics.

Clinical outcome measures

The omalizumab and placebo treated groups will be compared for changes in the following clinical outcomes (for repeated measurements such as daily peak flow and symptoms the mean values of the first and last 10 days of the relevant study period will be compared).

1. prior to reduction of existing anti-asthma therapy (first 12 weeks of study):

   * Pre-bronchodilator FEV1 (primary outcome measure)
   * Morning and evening peak expiratory flow
   * Exhaled nitric oxide
   * Day and night time symptom scores
   * Total dosages of rescue beta2-agonist
   * Total symptom free days
   * Validated asthma Quality of Life scores
2. during anti-asthma therapy reduction phase (subsequent 8 weeks of study):

   * The primary outcome measure will be disease exacerbation, defined as a need for rescue oral corticosteroid medication for worsening of symptoms and/or deterioration in lung function, as agreed between the patient and the study physician
   * Secondary outcome measures will include all those measurements listed in section (a) above, unless they cannot be measured because of disease exacerbation (the primary outcome measure)

Laboratory outcome measures

These will arise from immunological, immunohistochemical and molecular analysis of peripheral blood and bronchial biopsies taken from all patients at the beginning and end of the first 12 weeks of the study prior to reduction of anti-asthma therapy and will comprise of changes in:

* Lay down of collagen types I, III, IV and V and tenascin
* Vascular structures and angiogenic stimuli (collagen type IV, CD31 and human VEGF (29,30)
* Inflammatory cells (eosinophils, T cells, B cells, plasma cells, macrophages, neutrophils, mast cells)
* Goblet cells will be stained using monoclonal anti-Muc-5AC antibody
* Immunoglobulin E and its high- and low-affinity receptors will be stained using specific monoclonal antibodies as in our previous studies. B cells (CD20+) and plasma cells (CD138+) will be examined for expression of free kappa and lambda IgE light chains using double, sequential IHC.

Staining analysis: Entire areas of stained biopsy sections will be subjected to image analysis using a Zeiss Vision KS300 system allowing objective, unbiased digital image analysis using a powerful macro language .

Cytokine and chemokine concentrations in endobronchial tissue homogenates: These will be measured in homogenates of 2 biopsies by electrochemiluminescence using the SECTOR Imager 6000 and assay kits produced by Meso Scale Discovery. The MS6000 Human TH1/TH2 10-Plex Base Kit will be used to measure IFN-gamma, IL-1beta, IL-2, IL-4, IL-5, IL-10, IL-12p70, IL-13, TNF-alpha. The MS6000 Human Chemokine 9-Plex Base Kit will be used to measure Eotaxin, Eotaxin-3, IL-8, IP-10, MCP-1, MCP-4, MDC, MIP-1beta, TARC.

IgE synthesis: Two biopsies from each patient will be snap frozen in RNA later for subsequent analysis of expression of switch circle transcripts and IgE mature and germline mRNA as in our previous recent publication and cloning of C-epsilon H-chain genes to look for evidence of clonal expansion of B cells caused by B cell superantigens. Two biopsies will be

\homogenised for extraction of B cells for cloning and analysis of IgE production by antigen microarray.

Serum: Stored serum samples taken at the time of bronchoscopy will be analysed for complete antigen-specific IgE repertoire using microarray, and anti-Fc-epsilon-RI activity using an in vitro basophil degranulation assay.

ELIGIBILITY:
Inclusion criteria-

* Males and females aged 18 to 60 years inclusive.
* Moderate or severe non-atopic asthma as defined below treated with inhaled corticosteroids for at least 6 months.
* Daytime and nighttime symptoms at least 3 days per week in the last 3 months prior to screening visit(despite taking inhaled corticosteroids with or without beta-2-agonists or leukotriene blockers.
* Pre-bronchodilator FEV1 40-80% of the predicted; reversibility equal to or more than 12% in response to inhaled beta-2-agonists documented at any time within the past 2 years.
* Negative skin prick and/or in vitro IgE tests to a range of 12 common aeroallergens(pollens:grass, hazel, alder, birch; danders: cat, dog; dust mite: D.pteronyssinus, D.farinae; moulds: Cladosporium, Aspergillus, Alternaria).

Exclusion Criteria

* Smoking within the past year or total smoking history more than 0.5 pack years.
* Pregnant or lactating females or those at risk of pregnancy.
* Treatment with more than 2000 mcg/day beclometasone, 1600 mcg/day budesonide or 1000 mcg/day fluticasone by inhalation or regular systemic corticosteroid at screening.
* Hospitalization for asthma or exacerbation requiring systemic corticosteroid therapy within 3 months of the screening visit.
* History of life threatening asthma, defined as an asthma episode that required intubations and/or was associated with hypercapnia, respiratory arrest and/or hypoxic seizures.
* Patients in whom, in the opinion of the study investigators, omalizumab therapy might normally require precaution (history of autoimmune disease, renal or hepatic impairment, hyperimmunoglobulin E syndrome, allergic bronchopulmonary aspergillosis and diabetes mellitus)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Pre-bronchodilator FEV1 | before and after treatment with omalizumab for 16 weeks
  Prior to reduction of existing anti-asthma therapy (first 12 weeks of study):
  • Pre-bronchodilator FEV1 (primary outcome measure)
Disease exacerbation | From week 12 to week 20 of the study
  During anti-asthma therapy reduction phase (subsequent 8 weeks of study):
  The primary outcome measure during asthma therapy reduction phase will be disease exacerbation defined as a need for rescue oral corticosteroid medication for worsening of symptoms and/or deterioration in lung function, as agreed between the patient and the study physician

SECONDARY OUTCOMES:
Day and night time symptom scores | before and after treatment with omalizumab for 16 weeks
  These will be measured using standard Asthma Control Questionnaires(ACQ)
Morning and evening peakflows | before and after treatment with omalizumab for 16 weeks
Exhaled nitric oxide | before and after treatment with omalizumab for 16 weeks(from week 0 to week 16)
Total dosage of rescue beta-2-agonists | before and after treatment with omalizumab for 16 weeks(from week 0 to week 16)
Total symptom free days | before and after treatment with omalizumab for 16 weeks(from week 0 to week 16)
Quality of life scores | before and after treatment with omalizumab for 16 weeks(from week 0 to week 16)
Markers of airway remodelling and inflammation | before and after treatment with omalizumab for 16 weeks(from week 0 to week 16)
  These include- Collagen,tenascin,VEGF,CD31,inflammatory cells,goblet cells etc.
Local IgE synthesis in the bronchial mucosa and its expression | before and after treatment with omalizumab for 16 weeks(from week 0 to week 16)
  The measurement will include- IgE, its low and high affinity receptors, expression of free kappa and lambda light chains on B-cells and plasma cells

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Corrigan, MD, PhD, Principal Investigator — King's College, London, UK; Neil Barnes, MD, Principal Investigator — London Chest Hospital, UK; Prathap Pillai, MD, Principal Investigator — King's College London
Locations (2):
- United Kingdom (2):
  - London Chest Hospital, London
  - Guy's Hospital, London, UK, London

REFERENCES:
- [Derived] Pillai P, Chan YC, Wu SY, Ohm-Laursen L, Thomas C, Durham SR, Menzies-Gow A, Rajakulasingam RK, Ying S, Gould HJ, Corrigan CJ. Omalizumab reduces bronchial mucosal IgE and improves lung function in non-atopic asthma. Eur Respir J. 2016 Dec;48(6):1593-1601. doi: 10.1183/13993003.01501-2015. Epub 2016 Oct 20. PMID 27824606